CLINICAL TRIAL: NCT06350084
Title: The Effect of Mother's Touch and Nurse's Therapeutic Touch on Pain Level and Crying Time During Heel Blood Collection in Newborns: A Randomized Controlled Study
Brief Title: Effect of Mother's Touch and Nurse's Therapeutic Touch on Pain Level and Crying Time During Heel Blood Collection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Selda Ateş Beşirik, Principal Investigator, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/381
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Pain, Acute; Newborn; Crying
Keywords: Newborn; Pain; Therapeutic Touch; Touch; Heel Stick
MeSH Terms: conditions — Acute Pain; Crying; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mother's Touch Group (Experimental): Heel blood will be taken while the infant was Mother's Touch. Mother's touch will be applied to the infants before, during and after the procedure.
  Interventions: Behavioral: Mother's Touch
- Nurse's Therapeutic Touch Group (Experimental): Heel blood will be taken while the infant was Nurse's Therapeutic Touch.Therapeutic Touch will be applied to the infants before, during and after the procedure.
  Interventions: Behavioral: Nurse's Therapeutic Touch
- Control Group (No Intervention): In this group, infants received routine heel blood collection procedure.

INTERVENTIONS:
Behavioral: Mother's Touch — Heel blood will be taken while the infant was Mother's Touch. Mother's touch will be applied to the infants before, during and after the procedure.
  Arms: Mother's Touch Group
Behavioral: Nurse's Therapeutic Touch — Heel blood will be taken while the infant was Nurse's Therapeutic Touch.Therapeutic Touch will be applied to the infants before, during and after the procedure.
  Arms: Nurse's Therapeutic Touch Group

SUMMARY:
This prospective study is planned as a randomized controlled study with the purpose of determining the effect of Mother's Touch and Nurse's Therapeutic Touch on pain levels and crying times by newborns during heel blood collection.

DETAILED DESCRIPTION:
Among the non-pharmacological methods frequently used to reduce the effects of invasive interventions on the newborn; Practices such as reducing environmental stimuli, individualized developmental care, music therapy, breast milk, pacifier giving, sucrose, non-nutritive sucking, oral sucrose, kangaroo care, facilitated tucking position, and sweet solutions, massage and touching, positioning, nesting, kangaroo care, fetal positioning are included.

This study is a prospective, randomized and controlled trial. In this study aim, the effect of Mother's Touch and Nurse's Therapeutic Touch applied during heel blood collection on the pain levels and crying times in newborns will be examined.

Sample of the study consisted of a total of 120 newborns who met the sample selection criteria and were selected via randomization method. Newborns were divided into three groups; Mother's Touch group, Nurse's Therapeutic Touch group, and Control group.

Data were collected using the Infant-family Information Form, NIPS-Neonatal Infant Pain Scale, and Crying Follow-up Form.

ELIGIBILITY:
Inclusion Criteria:

* Parents who volunteered and gave consent to participate in the research
* Full term neonates (38-42 weeks of gestation)
* Underwent heel stick blood drawing for routine metabolic screening
* Aged 1 to 4 days
* Passed the hearing screening
* Birth weight between 2500-4400 grams
* Parents who know how to read, write and speak Turkish.

Exclusion Criteria:

* Parents with any mental problems
* Infants with any chronic disease and congenital anomalies.

Ages: 2 Days to 4 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
NIPS (Neonatal Infant Pain Scale) | during the heel blood collection procedures (10 minutes)
  It was developed in 1993 to evaluate interventional pain in newborns. Its Turkish adaptation was made in 1999. NIPS is an assessment tool that focuses on six behavioral responses of newborns: facial expressions, crying, breathing, arm movements, leg movements, and arousal. A score between 0 and 7 is obtained from the scale, and as the score obtained from the scale increases, the pain of newborns also increases. In the Turkish adaptation study of the scale, the Cronbach's alpha value was calculated as 0.83 before the procedure, 0.83 during the procedure and 0.86 after the procedure.

SECONDARY OUTCOMES:
Crying times | during the heel blood collection procedures (average 10 minutes)
  Duration of crying were recorded.
Processing time | during the heel blood collection procedures (average 10 minutes)
  Duration of heel blood collection procedure were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Selda Ateş Beşirik, PhD., Principal Investigator — Burdur Mehmet Akif Ersoy University; Emine Geçkil, Professor, Study Director — Necmettin Erbakan University
Locations (1):
- Burdur Bucak State Hospital, Burdur, Bucak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this study, after deidentification, will be shared with researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code